CLINICAL TRIAL: NCT01003184
Title: Efficacy of Once-Weekly Exenatide Versus Once or Twice Daily Insulin Detemir in Patients With Type 2 Diabetes Treated With Metformin Alone or in Combination With Sulphonylurea
Brief Title: Efficacy of Once-Weekly Exenatide Versus Once or Twice Daily Insulin Detemir in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-EW-GWDL
Record Dates: First submitted 2009-10-15; First posted 2009-10-28 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide once weekly; Byetta; insulin detemir; Levemir; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: exenatide once weekly
- 2 (Active Comparator)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, 2mg, once a week
  Arms: 1
Drug: insulin detemir — subcutaneous injection, with dosage titrated according to the determir label and published titration schedule, once or twice a day
  Other Names: Levemir
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effects of exenatide once weekly (QW) and insulin detemir with respect to glycemic control, body weight, lipids, safety, tolerability, and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have suboptimal glycaemic control as evidenced by an HbA1c 7.1% to 10.0%, inclusive
* Have a body mass index (BMI) of 25 kg/m2 to 45 kg/m2, inclusive
* Are receiving metformin at a stable dose (consistent with country specific requirements) of a minimum of 1000mg for at least 3 months prior to start start OR are receiving metformin at a minimum dose (consistent with country specific requirements) of 1000mg and sulphonylurea (as separate medications not as a fixed dose combination) at stable doses for 3 months prior to study start

Exclusion Criteria:

* Have any contraindication for the OAD that they have been using
* Have a known allergy or hypersensitivity to insulin detemir, exenatide or excipients contained in these agents
* Have been treated within 4 weeks of screening with systemic glucocorticoid therapy by oral, intravenous (IV) or intramuscular (IM) route, or are regularly treated with potent, inhaled intranasal steroids that are known to have a high rate of systemic absorption. Exceptions to this criterion include patients who are receiving glucocorticoid therapy for corticotropic hypopituitary deficiency (e.g. Addison disease)
* Have been treated with drugs that promote weight loss, within 3 months of screening
* Have been treated for longer than 2 weeks with any of the following excluded medications within 3 months prior to screening: insulin, alpha-glucosidase, Byetta® (exenatide BID formulation), thiazolidinediones (TZD), dipeptidyl peptidase (DPP)-4 inhibitors
* Have previously completed or withdrawn from this study or any other study investigating exenatide QW
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (34):
- Research Site, Dublin, Ireland
- United Kingdom (33):
  - Research Site, Addlestone, England
  - Research Site, Bath, England
  - Research Site, Birmingham, England
  - Research Site, Blackburn, England
  - Research Site, Bournemouth, England
  - Research Site, Chippenham, England
  - Research Site, Derby, England
  - Research Site, Exeter, England
  - Research Site, High Wycombe, England
  - Research Site, Hull, England
  - Research Site, Leicester, England
  - Research Site, Liverpool, England
  - Research Site, London, England
  - Research Site, Manchester, England
  - Research Site, Merseyside, England
  - Research Site, Middlesbrough, England
  - Research Site, Newcastle, England
  - Research Site, Northampton, England
  - Research Site, Oldham, England
  - Research Site, Plymouth, England
  - Research Site, Portsmouth, England
  - Research Site, Sheffield, England
  - Research Site, Stevenage, England
  - Research Site, Suffolk, England
  - Research Site, Wakefield, England
  - Research Site, Wiltshire, England
  - Research Site, Aberdeen, Scotland
  - Research Site, Dundee, Scotland
  - Research Site, Carmathen, Wales
  - Research Site, Swansea, Wales
  - Research Site, Wrexham, Wales
  - Research Site, Leytonstone
  - Research Site, Livingston

REFERENCES:
- [Derived] Guja C, Frias JP, Suchower L, Hardy E, Marr G, Sjostrom CD, Jabbour SA. Safety and Efficacy of Exenatide Once Weekly in Participants with Type 2 Diabetes and Stage 2/3 Chronic Kidney Disease. Diabetes Ther. 2020 Jul;11(7):1467-1480. doi: 10.1007/s13300-020-00815-z. Epub 2020 Apr 18. PMID 32306296

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 patients who were enrolled and randomized, subsequently discontinued the study before receiving study drug. These patients were not included in analysis.
Groups:
- Exenatide Once Weekly: Exenatide once weekly : subcutaneous injection, 2mg, once a week
- Insulin Detemir: Insulin detemir : subcutaneous injection, with dosage titrated according to the detemir label and published titration schedule, once or twice a day
Period: Overall Study
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Started | 111 | 111
Full Analysis Set (FAS) | 111 | 105
Completed | 92 | 99
Not Completed | 19 | 12
Not completed — Adverse Event | 12 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Loss of glucose control | 1 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly | Insulin Detemir | Total
Number analyzed (Participants) | 111 | 105 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 78 | 152
  >=65 years | 37 | 27 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.86) | 57.8 (9.48) | 58.5 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 33 | 73
  Male | 71 | 72 | 143
HbA1c [Mean (Standard Deviation); unit: Percentage of total hemoglobin] — At visit 3 (week 0).
  Percentage of total hemoglobin | 8.4 (0.85) | 8.4 (0.88) | 8.4 (0.86)
Weight [Mean (Standard Deviation); unit: Kilograms] | 96.7 (17.03) | 97.9 (15.82) | 97.3 (16.42)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Glycosylated Hemoglobin (HbA1c) Concentration ≤7.0% With Weight Loss (≥1.0 kg) at Endpoint (Week 26)
Description: The primary endpoint is the percentage of patients achieving HbA1c concentration ≤7.0% with weight loss (≥1.0 kg) at endpoint. The last post-baseline measurement set of both non-missing HbA1c concentration and weight (measured at the same time point, i.e. visit) is used as endpoint value. Patients who do not have a baseline weight measurement, have a protocol violation of baseline HbA1c <=7.0%, and/or have missing post-baseline measurements for HbA1c concentration and/or weight, are included in the analysis as non-responders regarding the primary objective.
Time Frame: Baseline, Week 26
Population: The full analysis set (FAS) includes all data from all randomised patients receiving at least one dose of the study drug according to the treatment the patients were assigned.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 111 | 105
Percentage | 44.1 [34.7 to 53.9] | 11.4 [6.0 to 19.1]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; Primary objective: to test hypothesis that the percentage of patients with HbA1c ≤7.0% with weight loss (≥1.0 kg) after exenatide QW is superior to insulin detemir. Sample size estimation: based on the test for difference in percentage between Exenatide QW and insulin detemir. Assuming: common drop-out rate 20%, response rate at endpoint 50% in the exenatide QW group and 25% in the insulin detemir group; 5% significance. 214 patients will provide 90% power to detect a difference; Test type: Superiority or Other; p < .0001, Regression, Logistic; Logistic regression model includes treatment group, use of SU (yes/no), baseline HbA1c and baseline weight as main factors; Odds Ratio (OR) = 6.60, 95% CI 2-sided [3.17 to 13.73]

2. Secondary Outcome: Percentage of Patients Who Have Achieved HbA1c ≤7.4% With Weight Loss (≥1.0 kg) at Endpoint (Week 26)
Description: Percentage of patients who have achieved HbA1c ≤7.4% with weight loss (≥1.0 kg) at endpoint (Week 26)
Time Frame: Baseline, Week 26
Population: The analysis was done for the FAS population (as randomised). For secondary analyses including both final HbA1c concentration and change in weight the last post-baseline measurement set of both non-missing HbA1c and weight was used as endpoint value.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 107 | 101
Percentage | 58.9 [49.0 to 68.3] | 17.8 [10.9 to 26.7]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; Test type: Superiority or Other; p < .0001, Regression, Logistic; Logistic regression model includes the independent variables treatment group, use of SU (yes/no), baseline HbA1c and baseline weight; Odds Ratio (OR) = 7.06, 95% CI 2-sided [3.64 to 13.70]

3. Secondary Outcome: Change in HbA1c From Baseline to Week 26
Description: Change in HbA1c from baseline to week 26
Time Frame: Baseline, Week 26
Population: The analysis was done for the FAS population (as randomised).
Measure: Least Squares Mean (Standard Error); unit: Percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 95 | 96
Percentage of total hemoglobin | -1.32 (0.076) | -0.91 (0.077)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; Mixed model repeated measures (MMRM) includes baseline value as covariate, study treatment, use of SU (yes/no), week of visit and treatment-by-week interaction as fixed effects and patient and error as random effects; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -0.41, 95% CI 2-sided [-0.62 to -0.20], Standard Error of Mean 0.104

4. Secondary Outcome: Change in Body Weight From Baseline to Week 26
Description: Change in body weight from baseline to week 26
Time Frame: Baseline, Week 26
Population: The analysis was done for the FAS population (as randomised).
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 96 | 98
kilograms | -2.79 (0.347) | 0.88 (0.351)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; Mixed model repeated measures MMRM) includes baseline value as covariate, study treatment, use of SU (yes/no), baseline HbA1c stratum, week of visit and treatment-by-week interaction as fixed effects and patient and error as random effects; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Least Squares Mean Difference = -3.67, 95% CI 2-sided [-4.63 to -2.71], Standard Error of Mean 0.488

5. Secondary Outcome: Percentage of Patients Achieving HbA1c ≤7.4% at Endpoint
Description: Percentage of patients who have achieved HbA1c ≤.7.4% at endpoint
Time Frame: Week 26
Population: The analysis was done for the FAS population (as randomised). Patients with baseline HbA1c ≤7.0% and/or no post-baseline HbA1c measurement were regarded as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 111 | 105
Percentage | 66.7 [57.1 to 75.3] | 54.3 [44.3 to 64.0]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; Logistic regression model includes independent variables treatment group, use of SU (yes/no), and baseline HbA1c; Test type: Superiority or Other; p = 0.0497, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.00 to 3.18]

6. Secondary Outcome: Percentage of Patients Achieving ≤7.0% at Endpoint
Description: Percentage of patients achieving ≤7.0% at endpoint.
Time Frame: Week 26
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 111 | 105
Percentage | 51.4 [41.7 to 61.0] | 34.3 [25.3 to 44.2]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; Logistic regression model includes independent variables treatment group, use of SU (yes/no), and baseline HbA1c; Test type: Superiority or Other; p = 0.0074, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.24 to 3.96]

7. Secondary Outcome: Percentage of Patients Achieving ≤6.5% at Endpoint
Description: Percentage of patients achieving HbA1c ≤6.5% at endpoint
Time Frame: Week 26
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 111 | 105
Percentage | 27.9 [19.8 to 37.2] | 7.6 [3.3 to 14.5]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; Logistic regression model includes independent variables treatment group, use of SU (yes/no), and baseline HbA1c; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 4.89, 95% CI 2-sided [2.10 to 11.35]

8. Secondary Outcome: Change in Fasting Serum Glucose From Baseline to Endpoint (Week 26).
Description: Change in fasting serum glucose from baseline to endpoint (Week 26).
Time Frame: Baseline, Week 26
Population: The analysis was done for the FAS population (as randomised).
  The last observation carried forward (LOCF) of post baseline values was used for this analysis.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 108 | 104
mmol/L | -2.33 (0.191) | -2.43 (0.196)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; ANCOVA model includes treatment group, baseline value, use of SU (yes/no) and baseline HbA1c stratum as factors; Test type: Superiority or Other; p = 0.6993, ANCOVA; Least Squares Mean Difference = 0.10, 95% CI 2-sided [-0.41 to 0.61], Standard Error of Mean 0.257

9. Secondary Outcome: Changes in Systolic Blood Pressure From Baseline to Week 26
Description: Change in systolic blood pressure from baseline to Week 26
Time Frame: Baseline, Week 26
Population: The analysis was done for the FAS population (as randomised).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 95 | 98
mmHg | -7.37 (1.342) | -2.65 (1.339)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; Mixed model repeated measures (MMRM) includes baseline value as covariate, study treatment, use of SU (yes/no), baseline HbA1c stratum, week of visit and treatment-by-week interaction as fixed effects and patient and error as random effects; Test type: Superiority or Other; p = 0.0116, Mixed Models Analysis; Least Squares Mean Difference = -4.72, 95% CI 2-sided [-8.37 to -1.07], Standard Error of Mean 1.853

10. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 26.
Description: Change in diastolic blood pressure from baseline to week 26.
Time Frame: Baseline, Week 26
Population: The analysis was done for the FAS population (as randomised).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 95 | 98
mmHg | -0.79 (0.855) [-1.79 to 0.56] | -0.34 (0.859) [-2.05 to 0.39]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.7034, Mixed Models Analysis; Least Squares Mean Difference = -0.45, 95% CI 2-sided [-2.77 to 1.88], Standard Error of Mean 1.179

11. Secondary Outcome: Change in Total Cholesterol From Baseline to Endpoint (Week 26).
Description: Change in total cholesterol from baseline to endpoint (week 26).
Time Frame: Baseline, Week 26
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 105 | 100
mmol/L | -0.09 (0.067) [-0.22 to 0.04] | 0.06 (0.068) [-0.08 to 0.19]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; ANCOVA model includes treatment group, baseline value, use of SU (yes/no) and baseline HbA1c stratum as factors; Test type: Superiority or Other; p = 0.1061, ANCOVA; Least Squares Mean Difference = -0.15, 95% CI 2-sided [-0.32 to 0.03], Standard Error of Mean 0.090

12. Secondary Outcome: Change in High-density Lipoprotein (HDL) Cholesterol From Baseline to Endpoint (Week 26).
Description: Change in High-density lipoprotein (HDL) cholesterol from baseline to endpoint (week 26).
Time Frame: Baseline, Week 26
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 105 | 100
mmol/L | 0.02 (0.014) [-0.01 to 0.05] | 0.04 (0.015) [0.01 to 0.06]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; ANCOVA model includes treatment group, baseline value, use of SU (yes/no) and baseline HbA1c stratum as factors; Test type: Superiority or Other; p = 0.4638, ANCOVA; Least Squares Mean Difference = -0.01, 95% CI 2-sided [-0.05 to 0.02], Standard Error of Mean 0.020

13. Secondary Outcome: Change in Triglycerides From Baseline to Endpoint (Week 26).
Description: Change in triglycerides from baseline to endpoint (week 26).
Time Frame: Baseline, Week 26
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 105 | 100
mmol/L | -0.01 (0.079) [-0.17 to 0.15] | -0.08 (0.081) [-0.24 to 0.08]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; ANCOVA model includes treatment group, baseline value, use of SU (yes/no) and baseline HbA1c stratum as factors; Test type: Superiority or Other; p = 0.4967, ANCOVA; Least Squares Mean Difference = 0.07, 95% CI 2-sided [-0.14 to 0.28], Standard Error of Mean 0.107

14. Secondary Outcome: Hypoglycemia Rate Per Year
Description: All confirmed hypoglycemia episodes defined as either minor (any time a patient feels that he or she is experiencing a sign or symptom associated with hypoglycaemia and blood glucose (BG) <3.0 mmol/L (54 mg/dL)) or major (any hypoglycaemic episode with symptoms consistent with hypoglycaemia, resulting in loss of consciousness or seizure, and shows prompt recovery in response to administration of glucagon or glucose, or BG measurement < 3.0mmol/L is available and the patient is not capable of self-treating were taken into account.
Time Frame: Baseline, Week 26
Population: Full analysis set (as randomized).
Measure: Number (95% Confidence Interval); unit: events per subject-year
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Number analyzed (Participants) | 111 | 105
events per subject-year | 0.06 [0.02 to 0.20] | 0.10 [0.03 to 0.30]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Detemir; The number of episodes by patient were compared between treatment groups using a poisson model with effects for treatment and baseline HbA1c and the logarithm of the days of exposure as the offset variable; Test type: Superiority or Other; p = 0.3247, Poisson regression; Ratio = 0.58, 95% CI 2-sided [0.19 to 1.72], Standard Error of Mean 0.322

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly | Insulin Detemir
Serious Adverse Events (participants affected / at risk) | 6/111 | 6/105
Other Adverse Events (participants affected / at risk) | 87/111 | 58/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=111) | Insulin Detemir (N=105)
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Blood amylase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal injury (Renal and urinary disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=111) | Insulin Detemir (N=105)
Nausea (Gastrointestinal disorders) | 53 | 12
Diarrhoea (Gastrointestinal disorders) | 19 | 11
Vomiting (Gastrointestinal disorders) | 16 | 9
Constipation (Gastrointestinal disorders) | 10 | 3
Dyspepsia (Gastrointestinal disorders) | 7 | 1
Injection site nodule (General disorders) | 22 | 0
Injection site pruritus (General disorders) | 12 | 1
Malaise (General disorders) | 6 | 2
Nasopharyngitis (Infections and infestations) | 23 | 31
Lower respiratory tract infection (Infections and infestations) | 5 | 6
Influenza (Infections and infestations) | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Headache (Nervous system disorders) | 23 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No